CLINICAL TRIAL: NCT02524990
Title: Simplified Medical Abortion Follow-Up Study
Brief Title: Simplified Medical Abortion Follow-Up
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Integrated into another study
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1024
Record Dates: First submitted 2015-08-11; First posted 2015-08-17 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Abortion; Pregnancy Tests
Keywords: Medical abortion; pregnancy tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Home-based follow-up with SQPT (Experimental): For the intervention, a semiquantitative pregnancy test (SQPT) will be performed at the health center before the participants take mifepristone, and again two weeks later by the participants, at home. Study staff will call the participants at two weeks to follow-up with the participants.
  Interventions: Behavioral: Home-based follow-up with SQPT

INTERVENTIONS:
Behavioral: Home-based follow-up with SQPT — Participants will be followed-up at home. They will receive an SQPT to perform at home two weeks after enrollment, and a scheduled follow-up phone call by study providers to determine the outcome of the procedure.
  Other Names: Simplified Medical Abortion Follow-Up Study

SUMMARY:
The purpose of this operations research study is to evaluate women's interest in and compliance with using a semiquantitative multi-level dipstick pregnancy test at home for medical abortion follow-up.

ELIGIBILITY:
Inclusion Criteria:

* She has been determined by the site investigator or designee to be fully eligible for medical abortion with mifepristone followed by misoprostol according to the site's standard criteria;
* She is willing to use the semiquantitative pregnancy test at home;
* She is wiling and able to comply with the study procedures;
* She speaks and reads English;
* She has signed the study informed consent form.

Ages: 11 Years to 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patients' compliance in performing the semiquantitative pregnancy test and reporting results | Within 2 weeks after medical abortion
  This will be assessed with a survey administered at the scheduled follow-up phone call. The survey will determine if the patient performed the SQPT as requested, and whether they can interpret and report the results correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, MD,MPH, Study Director — Gynuity Health Projects
Locations (1):
- Carafem Health Center, Chevy Chase, Maryland, United States